CLINICAL TRIAL: NCT00715910
Title: Long-term Antibody Persistence of GSK Biologicals' MenACWY-TT Vaccine Versus Menactra® in Healthy Adolescents/Adults Aged 10-25 Years and Booster Response to MenACWY-TT Vaccine Administered at 5 Years Post-primary Vaccination
Brief Title: The Long-term Antibody Persistence of GSK Biologicals' Meningococcal Vaccine GSK134612 in Healthy Adolescents/Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111670
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-09

CONDITIONS: Infections, Meningococcal
Keywords: Meningococcal vaccine; Booster vaccination; Immunogenicity; Meningococcal disease; Safety
MeSH Terms: conditions — Meningococcal Infections | interventions — tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine; Blood Specimen Collection

ARMS (6):
- Nimenrix 1 Group (Experimental): Subjects 11-25 years of age who were previously vaccinated with 1 dose of Nimenrix vaccine at the time of vaccination
  Interventions: Biological: Nimenrix; Procedure: Blood sampling
- Menactra Group (Active Comparator): Subjects 11-25 years of age who were previously vaccinated with 1 dose of Menactra vaccine at the time of vaccination
  Interventions: Biological: Nimenrix; Procedure: Blood sampling
- Nimenrix 2 Group (Experimental): Subjects 10<11 years of age who were previously vaccinated with 1 dose of Nimenrix vaccine at the time of vaccination
  Interventions: Biological: Nimenrix; Procedure: Blood sampling
- Nimenrix Naive Group (Experimental): Subjects 15 to <31 years of age at the time of primary vaccination with 1 dose of Nimenrix vaccine at year 5 of the current study
  Interventions: Biological: Nimenrix; Procedure: Blood sampling
- Nimenrix Pooled Group (Experimental): Pooled group of subjects 10-25 years of age from Nimenrix 1 and Nimenrix 2 groups in the primary study (NCT00454909) who had received 1 dose of Nimenrix vaccine in that study and will receive a booster dose in this current study.
  Interventions: Biological: Nimenrix
- Menactra Booster Group (Active Comparator): Subjects 11-25 years of age who had received 1 dose of Menactra vaccine in primary study (NCT00454909) and will receive 1 dose of Nimenrix vaccine in this current study.
  Interventions: Biological: Nimenrix

INTERVENTIONS:
Biological: Nimenrix — One dose, as intramuscular injection
  Other Names: Meningococcal vaccine GSK134612 (MenACWY-TT)
Procedure: Blood sampling — Blood samples will be collected from subjects 10-25 years of age as per enrollment in primary study and from subjects in the Nimerix Naive Group at Month 60 (Year 5) and 1 month post booster vaccination (Month 61).
  Arms: Menactra Group; Nimenrix 1 Group; Nimenrix 2 Group; Nimenrix Naive Group

SUMMARY:
In this study, the concentration of antibody to the vaccine one year, three and five years after vaccination in subjects who were vaccinated with GSK Biologicals' meningococcal vaccine GSK134612 and Menactra® in a previous study (whose objectives & outcome measures are presented in a separate protocol posting with NCT number =00454909) will be evaluated. The safety and immune response to a booster dose of vaccine GSK134612 administered at 5 years post-primary vaccination and a primary vaccination of a newly enrolled group with GSK 134612 vaccine will also be evaluated.

DETAILED DESCRIPTION:
GSK Biologicals has developed a meningococcal conjugate vaccine (GSK134612). This candidate vaccine has been shown to be well tolerated and immunogenic in subjects as of 12 months of age.

The purpose of this study is to evaluate the antibody persistence at approximately 1 year, 3 years and 5 years post-administration of one dose of GlaxoSmithKline (GSK) Biologicals' meningococcal vaccine GSK134612 as compared to Menactra® (meningococcal serogroups A, C, W-135 and Y-diphtheria toxoid conjugate vaccine, sanofi pasteur) when given to healthy adolescents/ adults 11 to 25 years of age In addition, the safety and immunogenicity of a booster dose of GSK134612 administered to all eligible subjects at 5 years after the primary vaccination will be evaluated.

Another cohort of subjects (naïve control group) 15 to <31 years of age will be offered a dose of MenACWY-TT vaccine at the same time to allow for evaluation of a primary (naïve control group) and booster dose within the same study.

This Protocol Posting has been updated following Protocol Amendment 1, May 2010 and Protocol Amendment 2, May 2011.

ELIGIBILITY:
Inclusion Criteria:

Persistence phase:

* A male or female who was between and including 10 and 25 years of age at the time of primary vaccination in the study with NCT number = 00454909.
* Written informed consent obtained from parents/guardian of the subject and written informed assent obtained from the subject if the subject is less than 18 years of age, or written informed consent obtained from the subject if the subject has achieved the 18th birthday.
* Healthy subjects as established by medical history.
* Having completed the active phase of the vaccination study with NCT number = 00454909.

Booster phase:

* Written informed consent obtained from parents/guardian of the subject and written informed assent obtained from the subject if the subject is less than 18 years of age, or written informed consent obtained from the subject if the subject has achieved the 18th birthday.
* Subjects who the investigator believes can and will comply with the requirements of the protocol should be enrolled in the study.
* Healthy subjects as established by medical history and history-directed physical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential, i.e., pre-menarche, have a current tubal ligation, hysterectomy, oophorectomy or be post-menopausal, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test on the day of vaccination and continue adequate contraception for 2 months after vaccination.

Additional inclusion criterion for the naïve control group:

• A male or female between, and including, 15 and 30 years of age at the time of the vaccination.

Exclusion Criteria:

Persistence phase:

* Use of any investigational or non-registered product within 30 days of each persistence time point.
* Vaccination with meningococcal polysaccharide or conjugate vaccine of serogroup A, C, W-135, and/or Y outside of study with NCT number = 00454909.
* History of any meningococcal disease due to serogroup A, B, C, W-135, or Y.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history.
* Administration of immunoglobulins and/or any blood products within the three months preceding each persistence time point.
* Concurrently participating in another clinical study within 30 days of each persistence time point, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy.
* Chronic alcohol or drug abuse.
* Subjects withdrew consent to be contacted for follow-up studies.

Booster phase (to be checked at Year 5 for all subject, including naïve control group):

* Child in care
* Not enrolled in the Kaiser Healthcare system.
* Use of any investigational or non-registered product within 30 days preceding administration of the study vaccine, or planned use throughout the extended safety follow-up period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior administration of the booster dose.
* Previous vaccination with meningococcal polysaccharide or conjugate vaccine of serogroup A, C, W-135, and/or Y outside of study with NCT number = 00454909.
* History of any meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition,including human immunodeficiency virus infection based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster vaccination or planned administration through Day 30 after vaccination.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy.
* History of chronic alcohol consumption and/or drug abuse.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting 30 days before until 30 days after the day of administration of the dose of vaccine(s) with the exception of any licensed inactivated influenza vaccine.
* Previous vaccination with tetanus and diphtheria toxoids within the last month.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of allergic disease or any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine, including latex.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Previous history of Guillain-Barré syndrome
* Acute disease at the time of vaccination.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 2 months after vaccination.
* For groups A, B and C only: Subjects withdrew consent to be contacted for follow-up studies.

Note: if the subject is female, prior to vaccination she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test on the day of vaccination and continue adequate contraception for 2 months after vaccination.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 818 (Actual)
Dates: Start 2008-07; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (9):
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fairfield, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Waianae, Hawaii
  - GSK Investigational Site, Waipio, Hawaii

REFERENCES:
- [Background] Baxter R et al. Immunogenicity and safety of an investigational quadrivalent meningococcal ACWY tetanus toxoid conjugate vaccine in healthy adolescents and young adults: 1-year follow-up. Abstract presented at the 51st Annual Interscience Conference on Antimicrobial Agents & Chemotherapy. Chicago, US, 17-20 September 2011.
- [Background] Baxter R et al. Antibody persistence and safety 3 years after a single dose of MenACWY-TT vaccine in healthy individuals aged 10-25 years. Abstract presented at the 31st Annual Meeting of European Society for Paediatric Infectious Diseases (ESPID), Milan, Italy, 28 May-1 June 2013.
- [Derived] Baxter R, Baine Y, Kolhe D, Baccarini CI, Miller JM, Van der Wielen M. Five-year Antibody Persistence and Booster Response to a Single Dose of Meningococcal A, C, W and Y Tetanus Toxoid Conjugate Vaccine in Adolescents and Young Adults: An Open, Randomized Trial. Pediatr Infect Dis J. 2015 Nov;34(11):1236-43. doi: 10.1097/INF.0000000000000866. PMID 26237742

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At Year 5, subjects in Nimenrix 1, Menactra and Nimenrix 2 groups received a booster dose of Nimenrix. During booster phase, subjects in Nimenrix 1 and Nimenrix 2 groups were pooled. An additional naïve control group 15 to < 31 years of age was enrolled at Year 5.
Pre-assignment Details: A total of 818 subjects were enrolled in the study. Year 1, 3 and 5 included only those subjects who came for the visits during these persistence years.
Groups:
- Nimenrix Pooled Group: Pooled group of subjects 10-25 years of age from Nimenrix 1 Group and Nimenrix 2 Group in the primary study (NCT00454909) who had received 1 dose of Nimenrix vaccine in that study and received a booster dose administered intramuscularly into the non-dominant deltoid in this current study during booster vaccination phase at Year 5.
- Menactra Booster Group: Subjects 11-25 years of age who had received 1 dose of Menactra vaccine in primary study (NCT00454909) and received 1 dose of Nimenrix vaccine administered intramuscularly into the non-dominant deltoid in this current study during booster vaccination phase at Year 5.
- Nimenrix Naïve Group: Naïve control group of subjects 15 to < 31 years at the time of primary vaccination with 1 dose of Nimenrix vaccine administered intramuscularly into the non-dominant deltoid in this current study during booster vaccination phase at Year 5.
Period: Year 1
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Started | 433 | 147 | 68 | 0 (Group not applicable during Year 1 Persistence phase) | 0 (Group not applicable during Year 1 Persistence phase) | 0 (Group not applicable during Year 1 Persistence phase)
Completed | 433 | 147 | 68 | 0 (Group not applicable during Year 1 Persistence phase) | 0 (Group not applicable during Year 1 Persistence phase) | 0 (Group not applicable during Year 1 Persistence phase)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Year 3
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Started | 345 | 86 | 56 | 0 (Group not applicable during Year 3 Persistence phase) | 0 (Group not applicable during Year 3 Persistence phase) | 0 (Group not applicable during Year 3 Persistence phase)
Completed | 345 | 86 | 56 | 0 (Group not applicable during Year 3 Persistence phase) | 0 (Group not applicable during Year 3 Persistence phase) | 0 (Group not applicable during Year 3 Persistence phase)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Year 5
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Started | 218 | 56 | 38 | 0 (Group not applicable during Year 5 Persistence phase) | 0 (Group not applicable during Year 5 Persistence phase) | 0 (Group not applicable during Year 5 Persistence phase)
Completed | 218 | 56 | 38 | 0 (Group not applicable during Year 5 Persistence phase) | 0 (Group not applicable during Year 5 Persistence phase) | 0 (Group not applicable during Year 5 Persistence phase)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Booster and ESFU Phase
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Started | 0 (Group not applicable during booster phase) | 0 (Group not applicable during booster phase) | 0 (Group not applicable during booster phase) | 183 | 38 | 101
Completed | 0 (Group not applicable during booster phase) | 0 (Group not applicable during booster phase) | 0 (Group not applicable during booster phase) | 172 | 36 | 88
Not Completed | 0 | 0 | 0 | 11 | 2 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 6 | 1 | 13
Not completed — Other | 0 | 0 | 0 | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of baseline subjects correspond to the subjects at Year 1 persistence phase and another cohort of subjects (naive control group) which was offered a dose of Nimenrix vaccine at Year 5 within the same study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group | Nimenrix naïve Group | Total
Number analyzed (Participants) | 433 | 147 | 68 | 101 | 749
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.9 (2.79) | 16.0 (2.83) | 11.2 (0.42) | 23.3 (4.74) | 16.5 (4.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 78 | 41 | 65 | 397
  Male | 220 | 69 | 27 | 36 | 352

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay (Using Human Complement) (hSBA) Titers Equal to or Above the Cut-off Values
Description: hSBA antibody titers were assessed for the hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY serogroups respectively. The antibody cut-off value assessed was equal to or above 1:8.
Time Frame: At year 1 persistence
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of persistence for Year 1, on all eligible subjects who had received primary vaccination during the primary study and who had available assay results for at least one tested antigen at the considered time point.
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 356 | 112 | 58
Subjects
  hSBA-MenA [N=350;111;57] | 102 | 35 | 15
  hSBA-MenC [N=336;105;56] | 319 | 77 | 55
  hSBA-MenW-135 [N=327;107;54] | 322 | 81 | 53
  hSBA-MenY [N=356;112;58] | 348 | 97 | 58

2. Primary Outcome: Number of Subjects With hSBA Titers Equal to or Above the Cut-off Values
Description: as for outcome 1
Time Frame: At year 3 persistence
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of persistence for Year 3, on all eligible subjects who had received primary vaccination during the primary study and who had available assay results for at least one tested antigen at the considered time point.
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 321 | 80 | 53
Subjects
  hSBA-MenA [N=314;78;51] | 117 | 37 | 22
  hSBA-MenC [N=317;80;53] | 295 | 65 | 51
  hSBA-MenW-135 [N=321;79;53] | 306 | 67 | 51
  hSBA-MenY [N=319;79;51] | 306 | 70 | 49

3. Primary Outcome: Number of Subjects With hSBA Titers Equal to or Above the Cut-off Values
Description: as for outcome 1
Time Frame: At year 5 persistence
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of persistence for Year 5, on all eligible subjects who had received primary vaccination during the primary study and who had available assay results for at least one tested antigen at the considered time point.
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 142 | 45 | 26
Subjects
  hSBA-MenA [N=141;45;24] | 69 | 20 | 9
  hSBA-MenC [N=140;44;26] | 130 | 35 | 22
  hSBA-MenW-135 [N=138;44;26] | 120 | 37 | 24
  hSBA-MenY [N=142;44;26] | 134 | 40 | 24

4. Secondary Outcome: Number of Subjects With hSBA Titers Equal to or Above the Cut-off Values
Description: hSBA antibody titers were assessed for the hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY serogroups respectively. The antibody cut-off value assessed was equal to or above 1:4.
Time Frame: At year 1 persistence
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 356 | 112 | 58
Subjects
  hSBA-MenA [N=350;111;57] | 106 | 35 | 17
  hSBA-MenC [N=336;105;56] | 319 | 77 | 55
  hSBA-MenW-135 [N=327;107;54] | 322 | 81 | 54
  hSBA-MenY [N=356;112;58] | 348 | 97 | 58

5. Secondary Outcome: Number of Subjects With hSBA Titers Equal to or Above the Cut-off Values
Description: as for outcome 4
Time Frame: At year 3 persistence
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 321 | 80 | 53
Subjects
  hSBA-MenA [N=314;78;51] | 123 | 37 | 23
  hSBA-MenC [N=317;80;53] | 295 | 68 | 51
  hSBA-MenW-135 [N=321;79;53] | 307 | 67 | 52
  hSBA-MenY [N=319;79;51] | 306 | 70 | 49

6. Secondary Outcome: Number of Subjects With hSBA Titers Equal to or Above the Cut-off Values
Description: as for outcome 4
Time Frame: At year 5 persistence
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 142 | 45 | 26
Subjects
  hSBA-MenA [N=141;45;24] | 74 | 20 | 9
  hSBA-MenC [N=140;44;26] | 134 | 39 | 24
  hSBA-MenW-135 [N=138;44;26] | 122 | 37 | 24
  hSBA-MenY [N=142;44;26] | 134 | 40 | 24

7. Secondary Outcome: hSBA Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) for the serogroups hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY respectively.
Time Frame: At year 1 persistence
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 356 | 112 | 58
Titers
  hSBA-MenA titers [N=350;111;57] | 5.4 [4.5 to 6.4] | 6.0 [4.3 to 8.5] | 5.2 [3.4 to 7.9]
  hSBA-MenC titers [N=336;105;56] | 172.0 [142.5 to 207.4] | 46.7 [30.2 to 72.1] | 238.3 [154.0 to 368.9]
  hSBA-MenW-135 titers [N=327;107;54] | 197.5 [173.0 to 225.5] | 48.9 [32.5 to 73.8] | 231.2 [174.5 to 306.2]
  hSBA-MenY titers [N=356;112;58] | 271.8 [237.5 to 311.2] | 100.8 [69.6 to 146.2] | 266.8 [205.1 to 347.0]

8. Secondary Outcome: hSBA Antibody Titers
Description: as for outcome 7
Time Frame: At year 3 persistence
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 321 | 80 | 53
Titers
  hSBA-MenA titers [N=314;78;51] | 6.2 [5.2 to 7.3] | 9.3 [6.2 to 14.0] | 8.8 [5.3 to 14.9]
  hSBA-MenC titers [N=317;80;53] | 117.9 [94.3 to 147.4] | 54.8 [33.9 to 88.9] | 131.2 [79.8 to 215.7]
  hSBA-MenW-135 titers [N=321;79;53] | 141.6 [122.8 to 163.4] | 75.5 [48.7 to 117.0] | 137.6 [98.2 to 192.9]
  hSBA-MenY titers [N=319;79;51] | 206.6 [177.9 to 239.8] | 139.0 [93.8 to 206.2] | 186.6 [130.7 to 266.6]

9. Secondary Outcome: hSBA Antibody Titers
Description: as for outcome 7
Time Frame: At year 5 persistence
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 142 | 45 | 26
Titers
  hSBA-MenA titers [N=141;45;24] | 8.9 [6.8 to 11.8] | 7.9 [4.8 to 13.2] | 6.3 [3.2 to 12.2]
  hSBA-MenC titers [N=140;44;26] | 94.6 [65.9 to 135.9] | 30.6 [17.3 to 54.4] | 92.9 [39.6 to 217.6]
  hSBA-MenW-135 titers [N=138;44;26] | 103.5 [76.3 to 140.5] | 70.4 [37.2 to 133.1] | 92.4 [50.5 to 168.8]
  hSBA-MenY titers [N=142;44;26] | 224.6 [173.9 to 290.0] | 129.3 [77.4 to 215.9] | 113.7 [58.4 to 221.3]

10. Secondary Outcome: Number of Subjects With Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSY, and Anti-PSW-135 Concentrations Equal to or Above the Cut-off Values
Description: The cut-off values were defined as a concentration ≥0.3 microgram per milliliter (μg/mL) and ≥2.0 μg/mL.
Time Frame: At year 1 persistence
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 366 | 112 | 59
Subjects
  Anti-PSA ≥ 0.3 µg/mL [N=355;112;56] | 340 | 101 | 55
  Anti-PSA ≥ 2.0 µg/mL [N=355;112;56] | 260 | 66 | 38
  Anti-PSC ≥ 0.3 µg/mL [N=366;112;58] | 302 | 56 | 51
  Anti-PSC ≥ 2.0 µg/mL [N=366;112;58] | 162 | 31 | 28
  Anti-PSW-135 ≥ 0.3 µg/mL [N=354;104;56] | 319 | 65 | 54
  Anti-PSW-135 ≥ 2.0 µg/mL [N=354;104;56] | 178 | 27 | 28
  Anti-PSY ≥ 0.3 µg/mL [N=358;112;59] | 342 | 78 | 55
  Anti-PSY ≥ 2.0 µg/mL [N=358;112;59] | 240 | 38 | 37

11. Secondary Outcome: Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSY, and Anti-PSW-135 Antibody Concentrations
Description: Antibody concentrations were given as geometric mean concentrations (GMCs) and expressed in μg/mL.
Time Frame: At year 1 persistence
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 366 | 112 | 59
μg/mL
  Anti-PSA [N=355;112;56] | 5.0 [4.2 to 5.9] | 3.7 [2.6 to 5.3] | 4.2 [2.9 to 6.1]
  Anti-PSC [N=366;112;58] | 1.8 [1.5 to 2.1] | 0.6 [0.5 to 0.9] | 2.1 [1.4 to 3.1]
  Anti-PSW-135 [N=354;104;56] | 2.0 [1.7 to 2.3] | 0.8 [0.6 to 1.1] | 2.0 [1.5 to 2.6]
  Anti-PSY [N=358;112;59] | 3.4 [3.0 to 4.0] | 1.0 [0.7 to 1.3] | 2.5 [1.8 to 3.4]

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Related to a Concurrent GSK Medication
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From 6 months up to 1 year following primary vaccination
Population: Analysis was performed on Total cohort at Year 1 which included all subjects vaccinated in the primary study and who came back to the visit at Year 1.
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 433 | 147 | 68
Subjects | 0 | 0 | 0

13. Secondary Outcome: Number of Subjects With SAEs Related to Study Participation or to a Concurrent GSK Medication
Description: as for outcome 12
Time Frame: From 6 months up to 3 years following primary vaccination
Population: Analysis was performed on Total cohort at Year 3 which included all subjects vaccinated in the primary study and who came back to the visit at Year 3.
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 345 | 86 | 56
Subjects | 0 | 0 | 0

14. Secondary Outcome: Number of Subjects With SAEs Related to Study Participation or to a Concurrent GSK Medication
Description: as for outcome 12
Time Frame: From 6 months up to 5 years following primary vaccination
Population: Analysis was performed on Total cohort at Year 5 which included all subjects vaccinated in the primary study and who came back to the visit at Year 5.
Measure: Number; unit: Subjects
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group
Number analyzed (Participants) | 218 | 56 | 38
Subjects | 0 | 0 | 0

15. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers Equal to or Above the Cut-off Values
Description: The cut-off values were defined as hSBA antibody titers ≥ 1:4 and ≥ 1:8.
Time Frame: 1 month post primary (naïve control group) and booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity at Month 61 which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after the primary (naïve control group) or booster vaccination.
Measure: Number; unit: Subjects
Groups:
- Nimenrix Naïve Group: Naïve control group of subjects 15 to <31 years at the time of primary vaccination with 1 dose of Nimenrix vaccine administered intramuscularly into the non-dominant deltoid in this current study during booster vaccination phase at Year 5
Arm/Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Number analyzed (Participants) | 109 | 29 | 84
Subjects
  hSBA-MenA ≥ 1:4 [N=106;28;79] | 105 | 28 | 61
  hSBA-MenA ≥ 1:8 [N=106;28;79] | 105 | 28 | 61
  hSBA-MenC ≥ 1:4 [N=109;29;81] | 108 | 29 | 78
  hSBA-MenC ≥ 1:8 [N=109;29;81] | 108 | 29 | 77
  hSBA-MenW-135 ≥ 1:4 [N=109;29;80] | 109 | 29 | 74
  hSBA-MenW-135 ≥ 1:8 [N=109;29;80] | 109 | 29 | 74
  hSBA-MenY ≥ 1:4 [N=109;29;84] | 109 | 29 | 82
  hSBA-MenY ≥ 1:8 [N=109;29;84] | 109 | 29 | 82

16. Secondary Outcome: hSBA Antibody Titers
Description: Titers are given as GMTs for the serogroups hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY respectively.
Time Frame: 1 month post primary (naïve control group) and booster vaccination
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Number analyzed (Participants) | 109 | 29 | 84
Titers
  hSBA-MenA Titers [N=106;28;79] | 783.8 [601.7 to 1020.9] | 952.0 [600.9 to 1508.2] | 79.7 [46.3 to 137.4]
  hSBA-MenC Titers [N=109;29;81] | 5020.4 [3995.4 to 6308.4] | 6722.1 [3950.9 to 11437.2] | 534.7 [308.0 to 928.1]
  hSBA-MenW-135 Titers [N=109;29;80] | 5517.6 [4573.6 to 6656.4] | 3729.0 [2415.4 to 5757.1] | 237.7 [150.4 to 375.8]
  hSBA-MenY Titers [N=109;29;84] | 5664.3 [4590.0 to 6990.1] | 6546.4 [4312.3 to 9938.0] | 755.1 [522.4 to 1091.4]

17. Secondary Outcome: Number of Subjects With Vaccine Response for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibodies
Description: Vaccine response was defined as:
  For initially seronegative subjects: antibody titre ≥ 1:8 at one month after vaccination For initially seropositive subjects: antibody titre at one month after vaccination ≥ 4 fold the titres before vaccination.
Time Frame: 1 month post primary (naïve control group) and booster vaccination
Population: as for outcome 15
Measure: Number; unit: Subjects
Arm/Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Number analyzed (Participants) | 106 | 29 | 78
Subjects
  hSBA-MenA [N=101;28;75] | 98 | 24 | 51
  hSBA-MenC [N=106;28;68] | 97 | 27 | 47
  hSBA-MenW-135 [N=105;28;76] | 101 | 24 | 51
  hSBA-MenY [N=106;29;78] | 97 | 27 | 53

18. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as occurrence of any solicited local symptom reported irrespective of intensity grade. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness and swelling were defined as redness/swelling above 50 millimeter (mm).
Time Frame: During the 4-day (Days 0-3) post primary (naïve control group) and booster vaccination
Population: Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects in the primary study with a booster vaccine administration documented, newly enrolled group administered primary vaccination at Year 5 and also had symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Number analyzed (Participants) | 170 | 37 | 91
Subjects
  Any Pain | 100 | 20 | 55
  Grade 3 Pain | 6 | 0 | 1
  Any Redness | 39 | 6 | 17
  Grade 3 Redness | 0 | 0 | 0
  Any Swelling | 27 | 5 | 14
  Grade 3 Swelling | 2 | 1 | 2

19. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms (nausea, vomiting, diarrhea and/or abdominal pain), headache and temperature. Any = occurrence of any general symptoms reported irrespective of intensity grade and relationship to study vaccination. Any temperature = axillary temperature greater than or equal to (≥)37.5 degrees Celsius (°C). Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 temperature = axillary temperature above 39.0°C. Related = symptoms considered by the investigator to have a causal relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) post primary (naïve control group) and booster vaccination
Population: as for outcome 18
Measure: Number; unit: Subjects
Arm/Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Number analyzed (Participants) | 170 | 37 | 91
Subjects
  Any Fatigue | 58 | 7 | 30
  Grade 3 Fatigue | 3 | 0 | 1
  Related Fatigue | 57 | 6 | 29
  Any Gastrointestinal symptoms | 28 | 8 | 20
  Grade 3 Gastrointestinal symptoms | 0 | 0 | 2
  Related Gastrointestinal symptoms | 28 | 8 | 17
  Any Headache | 61 | 10 | 22
  Grade 3 Headache | 0 | 0 | 1
  Related Headache | 60 | 10 | 21
  Any Temperature | 4 | 0 | 3
  Grade 3 Temperature | 0 | 0 | 0
  Related Temperature | 2 | 0 | 2

20. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Days 0-30) following primary (naïve control group) and booster vaccination
Population: as for outcome 18
Measure: Number; unit: Subjects
Arm/Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Number analyzed (Participants) | 183 | 38 | 101
Subjects | 40 | 9 | 16

21. Secondary Outcome: Number of Subjects Reporting New Onset Chronic Illness(es) (NOCIs)
Description: Examples of NOCIs include autoimmune disorders, asthma, type 1 diabetes and allergies.
Time Frame: During the 6-month period following the primary (naïve control group) and booster vaccination
Population: as for outcome 18
Measure: Number; unit: Subjects
Arm/Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Number analyzed (Participants) | 183 | 38 | 101
Subjects | 0 | 0 | 0

22. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 12
Time Frame: During the 6-month period following the primary (naïve control group) and booster vaccination
Population: as for outcome 18
Measure: Number; unit: Subjects
Arm/Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Number analyzed (Participants) | 183 | 38 | 101
Subjects | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs = From 6 months up to 5 years after primary vaccination and up to 6 months after vaccination in booster phase. Solicited and unsolicited symptoms during 4 days (Days 0-3) and 31-days (Days 0-30) after vaccination in booster phase respectively.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | Nimenrix 1 Group | Menactra Group | Nimenrix 2 Group | Nimenrix Pooled Group | Menactra Booster Group | Nimenrix Naïve Group
Serious Adverse Events (participants affected / at risk) | 0/433 | 0/147 | 0/68 | 3/183 | 0/38 | 0/101
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 100/183 | 20/38 | 55/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix 1 Group (N=433) | Menactra Group (N=147) | Nimenrix 2 Group (N=68) | Nimenrix Pooled Group (N=183) | Menactra Booster Group (N=38) | Nimenrix Naïve Group (N=101)
Appendicitis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 — Assessed during the 6 months period following vaccination in booster phase
Depression (Psychiatric disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 — Assessed during the 6 months period following vaccination in booster phase
Malaria (Infections and infestations) | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 — Assessed during the 6 months period following vaccination in booster phase
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix 1 Group (N=0) | Menactra Group (N=0) | Nimenrix 2 Group (N=0) | Nimenrix Pooled Group (N=183) | Menactra Booster Group (N=38) | Nimenrix Naïve Group (N=101)
Pain (General disorders) | 0 | 0 | 0 | 100/170 | 20/37 | 55/91 — Assessed during the 6 months period following vaccination in booster phase
Redness (General disorders) | 0 | 0 | 0 | 39/170 | 6/37 | 17/91 — Assessed during the 6 months period following vaccination in booster phase
Swelling (General disorders) | 0 | 0 | 0 | 27/170 | 5/37 | 14/91 — Assessed during the 6 months period following vaccination in booster phase
Fatigue (General disorders) | 0 | 0 | 0 | 58/170 | 7/37 | 30/91 — Assessed during the 6 months period following vaccination in booster phase
Gastrointestinal symptoms (General disorders) | 0 | 0 | 0 | 28/170 | 8/37 | 20/91 — Assessed during the 6 months period following vaccination in booster phase
Headache (General disorders) | 0 | 0 | 0 | 61/170 | 10/37 | 22/91 — Assessed during the 6 months period following vaccination in booster phase
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 0 — Assessed during the 6 months period following vaccination in booster phase

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.